CLINICAL TRIAL: NCT02447861
Title: The 3q29 Deletion and 3q29 Duplication: Architecture of Behavioral Phenotypes
Status: Recruiting | Type: Observational
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Jennifer Gladys Mulle, MHS, PhD, Associate Professor, Rutgers, The State University of New Jersey
Other Study IDs: Pro2021001976
Record Dates: First submitted 2015-05-15; First posted 2015-05-19 (Estimated); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Microdeletion 3q29 Syndrome; Microduplication 3q29 Syndrome
MeSH Terms: conditions — Chromosome 3q29 Deletion Syndrome; Chromosome 3q29 Duplication Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — DNA from saliva will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 3q29 deletion: Individuals with 3q29 deletion syndrome (sometimes called "3q29 micro deletion")
- 3q29 duplication: Individuals with 3q29 duplication syndrome (sometimes called "3q29 micro duplication")
- Parents: parents of individuals with the 3q29 deletion or 3q29 duplication
- Healthy Controls: Unrelated age-matched controls without 3q29 deletion or duplication

SUMMARY:
The 3q29 deletion syndrome is caused by a deletion of a small part of human chromosome 3, and the duplication syndrome is caused by a duplication of this same small region. The purpose of this study is to understand the medical and behavioral consequences of these syndromes.

DETAILED DESCRIPTION:
People with 3q29 deletion syndrome are missing a small part of a region on human chromosome 3, and people with 3q29 duplication syndrome have an extra part of their chromosome 3. Sometimes babies are born with a deletion or duplication of part of human chromosome 3, even though their parents have an intact chromosome 3. This is called de novo (or new) abnormalities.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of 3q29 deletion or 3q29 duplication
* Consent from parents or guardians or an adult with 3q29 deletion or 3q29 duplication that does not require a legal guardian or an adult who is the healthy sibling of an individual with 3q29 deletion or 3q29 duplication or a healthy age-matched control

Exclusion Criteria:

* Clinically significant medical disease that would prohibit participation in the study procedures

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study subjects will be recruited by an internet-based registry. The registry website will be indexed on popular search enginesand potential study subjects can elect to visit the website as they choose. Study population will be individuals with the 3q29 deletion or 3q29 duplication and their family members, although in most cases the primary caregiver of the 3q29 deletion or duplication individual will contribute the data. This study aims to collect data on approximately 200 individuals with the 3q29 deletion and 100 individuals with the 3q29 duplication. For comparison purposes, the study will assess an equal number of matched number of unaffected siblings and control individuals without the 3q29 deletion or duplication.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2013-07 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Range of medical conditions associated with the 3q29 deletion and duplication, assessed by the percent of patients reporting specific conditions present | 5 years
  A medical questionnaire designed to collect data on commonly reported medical conditions associated with the 3q29 deletion or duplication will be administered.

SECONDARY OUTCOMES:
T-score on the Behavior Rating Inventory of Executive Function (BRIEF) | Baseline, 5 years
  The BRIEF is a questionnaire designed to assess executive functioning. It is scored on a T-score scale, where higher scores indicate more disability in this domain. Scores range from 0-100.
Score on the Social Responsiveness Scale (SRS) | Baseline, 5 years
  The SRS is a 65-item, caregiver-rated assessment scale that measures observable items on social behavior and social language use, as well as characteristics of autism in a naturalistic social setting. Each item is rated on a scale from 0 (never true) to 3 (almost always true). The SRS total raw score ranges from 0 to 195; a higher score indicates greater severity of social impairment.
Score on the Social Communication Questionnaire (SCQ) | Baseline, 5 years
  The SCQ is a 40-item, parent-reported screening measure that taps the symptomatology associated with autism spectrum disorder (ASD). The items are in a yes/no format and are translated to scores of 1 (yes) or 0 (no). The threshold reflecting the need for diagnostic assessment is a score of 15. Higher scores are indicative of autism characteristics.
Score on the Child Behavior Checklist (CBCL) | Baseline, 5 years
  The CBCL is a 120-item, parent-reported checklist that includes several competence items, open-ended items for describing the child's illnesses, disabilities, concerns about the child, best things about the child, and several items to rate behavioral, emotional, and social problems. Responses are recorded on a Likert scale: 0 = Not True, 1 = Somewhat or Sometimes True, 2 = Very True or Often True. The standardized score is computed by determining the z-score by subtracting the mean for the subject's age group and gender from the raw score and then dividing this by the standard deviation for the subject's age group and gender. Next, multiply the z-score by 15 and then add 100. For activities scale, social scale, school scale, and total competence scale, higher values indicate higher competencies. For Internalizing problems, externalizing problems, and total problems, higher values indicate more problems.
Performance on the Penn Computerized Neurobahavioral Test battery (PennCNB) | Baseline, 5 years
  The PennCNB is a computerized assessment of domains of cognitive ability. It is scored on a z-score scale, where the mean is 0, positive scores indicate scores above the mean (better performance) and negative scores are below the mean (worse performance). Most acres wil fall between -3 and 3.
Prodromal Questionnaire - Brief Version (PQ-B) | Baseline, 5 years
  The PQ-B is a 21-item self-report screening measure for psychosis risk syndromes. Each item is rated on a five-point Likert scale from 1 (strongly disagree) to 5 (strongly agree). The total score ranges from 0 to 21, where respondents receive 1 point for each "yes" response. The threshold reflecting the need for diagnostic assessment is a score of 3 or higher.
Feeding questionnaire | Baseline
  Feeding questionnaire is an 11-item questionnaire to document the specific feeding problems experienced by individuals with 3q29 deletion syndrome.
Structured Interview for Psychosis Risk Syndromes (SIPS) | Baseline
  The Structured Interview for Psychosis Risk Syndromes (SIPS) is a semi-structured interview designed to assess early signs of psychosis. For each scale scores range from 0-6, with higher scores indicating worse performance
Score on the Vineland | 5 years
  The Vineland is a questionnaire designed to assess adaptive behavior. It is scores on a standard scale, where scores range from 0-160 with arena of 100. Higher scores indicated petter performance.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Mulle, MHS, PhD, Principal Investigator — Rutgers University
Locations (1):
- Internet-Based, Piscataway, New Jersey, United States

DOCUMENTS (1):
  • Informed Consent Form (2024-09-28): https://cdn.clinicaltrials.gov/large-docs/61/NCT02447861/ICF_000.pdf